CLINICAL TRIAL: NCT01437904
Title: A Pilot Study Assessing The Feasibility Of Outpatient Tubeless Percutaneous Nephrolithotomy (PCNL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Darren Beiko, Principal Investigator and Associate Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PCNL Beiko
Record Dates: First submitted 2011-09-20; First posted 2011-09-21 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Renal Calculi
Keywords: Renal Calculi; Percutaneous nephrolithotomy (PCNL)
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outpatient (Experimental): Outpatient recovery following Percutaneous nephrolithotomy
  Interventions: Procedure: Outpatient Recovery
- In hospital (Sham Comparator): Inpatient recovery following Percutaneous nephrolithotomy
  Interventions: Procedure: In hospital recovery

INTERVENTIONS:
Procedure: Outpatient Recovery — Patients go home following Percutaneous nephrolithotomy
  Arms: Outpatient
Procedure: In hospital recovery — Patients are hospitalized following Percutaneous nephrolithotomy
  Arms: In hospital

SUMMARY:
Outpatient tubeless Percutaneous nephrolithotomy (PCNL) could potentially improve patient care and result in significant cost savings for our hospital each year. If this pilot study is successful, Queen's/KGH will lead a collaborative national multicentre trial to further establish the role of this new approach in the surgical treatment of kidney stones.

DETAILED DESCRIPTION:
One in eight human beings will develop kidney stones during their lifetime. Percutaneous nephrolithotomy (PCNL) is the standard minimally invasive surgical operation for the removal of large kidney stones. Around the world, patients are routinely admitted to hospital following PCNL. The reasons that outpatient PCNL has not been otherwise attempted are related to the risk of bleeding and the need for an indwelling kidney drainage tube. Other than a single publication from the mid-1980's, there have been no other publications regarding outpatient PCNL up until this year, both from our group at Queen's University. We challenge the need for hospitalization following PCNL provided that proper technique for percutaneous renal access is used and patients are very carefully selected. In fact, we have safely performed outpatient tubeless PCNL on over 5 patients to date and we have two related published abstracts that were presented in 2008 at international Urology conferences in Albuquerque, New Mexico and Shanghai, China. Our manuscript titled "Totally tubeless outpatient percutaneous nephrolithotomy: initial case report" has been published in Advances in Urology in 2009. Additionally, a second manuscript of ours titled "Outpatient tubeless PCNL: the initial case series" is currently in press in the Canadian Urological Association Journal.

Outpatient PCNL offers patients several potential benefits, including decreased pain due to lack of nephrostomy tube, earlier and faster convalescence and lower rate of hospital acquired infections and complications. Furthermore, outpatient PCNL may offer several potential cost savings to the hospital and health care system, including the daily cost of an inpatient hospital bed, the imaging and procedural costs of antegrade nephrostogram, including the interventional radiologist's fee, the cost of nursing staff and the cost of intravenous antibiotics and other medications required by the hospitalized patient. Conversely, outpatient PCNL could potentially result in additional costs if emergency visits, readmissions and further interventions occur.

Project Synopsis This project is a pilot study that examines the safety, efficacy, feasibility and potential cost savings of performing percutaneous nephrolithotomy (PCNL) on an outpatient basis. If shown to be feasible, outpatient PCNL could result in significant potential cost savings to the hospital and health care system, as normal care following PCNL involves a 1-3 day hospital stay. The main objective of this pilot study is to obtain preliminary data necessary to develop a definitive national multicentre prospective randomized controlled trial comparing outpatient PCNL to standard PCNL.

Hypotheses Patients can be successfully randomized to outpatient versus standard PCNL and that outpatient PCNL will be a successful procedure.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for Percutaneous nephrolithotomy (PCNL) of renal calculi
* patient has normal renal function
* patient is 18 or older
* patient agrees to return for follow up
* ASA class 1 or 2

Exclusion Criteria:

* patient has had previous PCNL for same stone
* patient is pregnant
* patient would not be appropriate as participant (investigator's opinion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To randomize and successfully treat patients with outpatient PCNL versus standard PCNL. | One month
  To randomize and successfully treat patients with outpatient PCNL versus standard PCNL.

SECONDARY OUTCOMES:
Is there is a difference in costs, complications and stone-free rates between the two groups. | One month
  Is there a difference in costs, complications and stone-free rates between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Beiko, MD FRCSC, Principal Investigator — Queen's University
Locations (1):
- Centre for Applied Urological Research/Kingston General Hospital, Kingston, Ontario, Canada